CLINICAL TRIAL: NCT01389336
Title: Kontrollierte Klinische Nicht-randomisierte Pilotstudie Zur Komplexen Āyurveda-Therapie Beim Fibromyalgiesyndrom im Vergleich Zur Konventionellen Standardbehandlung
Brief Title: Add-on Complex Ayurvedic Treatment in Fibromyalgia-Syndrome Compared to Standard Care Alone
Acronym: KAFA
Status: Completed | Type: Observational
Sponsor: Andreas Michalsen (Other)
Collaborators: Dr.Heinz Horst Deichmann Foundation,Essen,Germany (Unknown)
Responsible Party: Sponsor-Investigator, Andreas Michalsen, Prof. Dr. Andreas Michalsen, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Other Study IDs: KAFA
Record Dates: First submitted 2011-07-06; First posted 2011-07-08 (Estimated); Last update posted 2013-05-08 (Estimated); Status verified 2013-05

CONDITIONS: Fibromyalgia Syndrome
Keywords: Fibromyalgia Syndrome; Fibromyalgia; Ayurveda; Traditional Indian Medicine; CAM; Pain; Chronic Widespread Pain
MeSH Terms: conditions — Fibromyalgia; Pain; Chronic Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Add-on Ayurveda - Group: In the Āyurveda add-on-group 20 patients will receive individualized treatment according to the Āyurveda diagnosis which may include manual treatments, massages, dietary advice, specific consideration of selected food items, āyurvedic lifestyle & yoga posture advice and daily self-applied massage on top of standard care.
- Standard Care: 20 Patients will receive the individually adjusted complex conventional standard care according to the current AWMF-guidelines including physiotherapy, occupational therapy, specific pain therapy and psychotherapy.

SUMMARY:
The aim of this study is to evaluate the effectiveness of an additive complex āyurvedic diagnosis and treatment compared to conventional standard care alone in stationary patients with Fibromyalgia Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* age between 18 and 70 years
* FMS according to current guidelines

Exclusion Criteria:

* change of pharmacological FMS treatment >= 6 weeks before inclusion
* pregnancy or breat feeding
* acute psychiatric condition
* severe acute somatic disease
* severechronic comorbidity
* obesity WHO >= II degree
* bloodcoagulation-disease
* intake of opiods
* current treatment with hyperthermia
* simultaneous participant in other trial
* praticipation in other trial during 6 month before inclusion

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and Women with Fibromyalgia-Syndrome between 18 und 70 years of age
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2011-07; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Fibromyalgia Impact Questionnaire (FIQ) | max. 3 weeks
  Change in FIQ after completion of IPD-treatment

SECONDARY OUTCOMES:
Functional Hanover Questionnaire (FFBH) | max. 3 weeks
State Trait Anxiety Inventory (STAI) | max. 3 weeks
Profile of Mood States (POMS) | max. 3 weeks
Short Form 36 Health Survey (SF-36) | max. 3 weeks
VAS for pain | max 3 weeks
Likert-Scales | max 3 weeks
FIQ | 6 month
FFBH, STAI, POMS, SF-36, VAS, Likert-Scales. | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Michalsen, Prof. Dr., Principal Investigator — Charité Medical University Berlin Germany
Locations (1):
- Immanuel Hospital Berlin, Berlin, State of Berlin, Germany

REFERENCES:
- [Derived] Kessler CS, Ostermann T, Meier L, Stapelfeldt E, Schutte S, Duda J, Michalsen A. Additive Complex Ayurvedic Treatment in Patients with Fibromyalgia Syndrome Compared to Conventional Standard Care Alone: A Nonrandomized Controlled Clinical Pilot Study (KAFA Trial). Evid Based Complement Alternat Med. 2013;2013:751403. doi: 10.1155/2013/751403. Epub 2013 Sep 1. PMID 24073008
- See also: Hospital Website — http://www.immanuel.de
- See also: University Website — http://www.charite.de